CLINICAL TRIAL: NCT03705598
Title: Tai Chi Intervention for Geriatric Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Tongjian You, Professor, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 297908
Record Dates: First submitted 2018-05-23; First posted 2018-10-15 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain; Falls
MeSH Terms: conditions — Chronic Pain | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light physical exercise (Placebo Comparator): Usual-pace walking, strength exercise, stretching exercise, and balance exercise.
  Interventions: Behavioral: Light physical exercise
- Tai Chi (Active Comparator): Tai Chi walking drills and Yang-style Tai Chi 8 forms.
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Light physical exercise — One hour each session, two sessions each week, for 24 weeks. Each session will be structured into three 15-minute segments (including warm-up activities/balance exercise/walking, upper and lower body strength exercise/walking, and stretching exercise/balance exercise/walking, respectively), each ending with a short break to record the Borg Rating of Perceived Exertion (RPE), followed by a 5-minute break time or cool-down/wrap-up session. The session will be taught by a certified exercise physiologist and a research assistant.
  Arms: Light physical exercise
Behavioral: Tai Chi — One hour each session, two sessions each week, for 24 weeks. Each session will be structured into three 15-minute segments (including warm-up activities/balance exercise/breathing exercise, Tai Chi walking drills, and Tai Chi 8-form, respectively), each ending with a short break to record the RPE, and followed by a 5-minute break or cool-down/wrap-up session. The session will be taught by an experienced Tai Chi instructor and a research assistant.
  Arms: Tai Chi

SUMMARY:
Accumulating evidence supports that more pain, whether measured by number of pain sites or pain severity, is associated with poorer cognitive function and mobility, and fall risk in older persons. Tai Chi which holistically integrates physical and cognitive functions offers the possibility not only of alleviating pain but also improving attention and mobility in the many older adults who have chronic multisite pain. This proposed full-size randomized controlled Tai Chi trial is a direct extension of the investigators' previous work examining chronic pain, attention demands, mobility and falls in the older population, and is built on the investigators' National Institute on Aging-supported Tai Chi feasibility and acceptability pilot studies among older adults with multisite pain and risk for falls. The goal of this single-blinded randomized controlled trial is to examine the effects of a 24-week Tai Chi intervention on chronic pain, cognition, mobility, fear of falling, and fall rate in older adults with multisite pain and at risk for falls. The results of this study will provide a foundation to establish the clinical significance of Tai Chi in the management of chronic multisite pain and to explore the mechanisms through which Tai Chi improves chronic pain symptoms and lowers fall rate in at-risk older adults.

DETAILED DESCRIPTION:
The investigators will measure pain severity, pain interference, and fear of falling at baseline, mid-point (3-month), and post-intervention (6-month), as well as rate of falls during the intervention (0- to 6-month) and the 6-month follow-up period (month 6 to month 12) in 266 older adults (Tai Chi: N=133, and light physical exercise control: N=133). In addition, they will measure pain-related biomarkers, cognition, single-task and dual-task gait function, free-living physical activity, and sleep at baseline, mid-point, and post-intervention. The primary aims are: 1. to examine the effects of Tai Chi on pain symptoms in older adults with multisite pain. It is hypothesized that older adults in the Tai Chi intervention will have less pain, measured as pain severity and interference, than those in the light physical exercise control group; 2. to examine the effects of Tai Chi on fear of falling and rate of falls in older adults with multisite pain. It is hypothesized that older adults in the Tai Chi intervention will have less fear of falling and fewer falls than those in the light physical exercise control group. The secondary/exploratory aims are: 3. to examine the effects of Tai Chi on pain-related biomarkers in older adults with multisite pain. It is hypothesized that Tai Chi intervention will have greater reductions in levels of pain-related biomarkers and and beta endorphin, than those in the light physical exercise control group; 4. to examine the roles of changes in pain symptoms in the change of fall rate by Tai Chi in older adults with multisite pain. It is hypothesized that the effect of Tai Chi on the reduced fall rate will be explained in part by improvements in pain symptoms in older adults with multisite pain; 5. to examine the roles of changes in cognition and cognitive motor function in the change of fall rate by Tai Chi in older adults with multisite pain. It is hypothesized that the reduced fall rate in the Tai Chi group will be mediated by changes in cognition and cognitive-motor function in older adults with multisite pain.

ELIGIBILITY:
Inclusion Criteria:

1. be 65 years or older
2. report chronic multisite (≥2 sites) musculoskeletal pain
3. have had 1 or more falls in the past year or current use of an assistive device (a cane or walker)
4. be able to walk 20 feet without help
5. be able to communicate in English

Exclusion Criteria:

1. actively engage in moderate to vigorous exercise for more than 40 min/week
2. practiced Tai Chi or other mind-body exercise within the past year, or practiced Tai Chi or other mind-body exercise regularly for at least 3 months within the past 5 years
3. have moderate to severe cognitive impairment (Mini-Mental State Examination (MMSE) score <18)
4. have a diagnosis of a disease/condition that would interfere with their study participation (e.g., rheumatoid arthritis, stroke, Parkinson's disease, degenerative neuromuscular disease, unstable cardiac disease, Alzheimer's disease or other dementia, terminal disease)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 24 weeks
  Pain severity will be assessed using the Brief Pain Inventory.
Pain interference | 24 weeks
  Pain interference will be assessed using the Brief Pain Inventory.
Fear of falling | 24 weeks
  Fear of falling will be assessed using the Tinetti Falls Efficacy Scale.
Rate of falls | 48 weeks
  Rate of falls will be assessed using monthly falls calendar postcards.

SECONDARY OUTCOMES:
C-reactive protein | 24 weeks
  Plasma levels of C-reactive protein will be measured using enzyme-linked immunosorbent assays.
Interleukin 6 | 24 weeks
  Plasma levels of interleukin 6 will be measured using enzyme-linked immunosorbent assays.
Tumor necrosis factor alpha | 24 weeks
  Plasma levels of tumor necrosis factor alpha will be measured using enzyme-linked immunosorbent assays.
Nuclear factor kappa B | 24 weeks
  Plasma levels of nuclear factor kappa B will be measured using enzyme-linked immunosorbent assays.
Beta endorphin | 24 weeks
  Plasma levels of beta endorphin will be measured using an enzyme-linked immunosorbent assay.
Attention | 24 weeks
  Attention will be assessed by using 4 subscales of the Test of Everyday Attention.
Executive function | 24 weeks
  Executive function will be assessed using the Trailmaking test, which requires the connection of sequentially numbered circles (part A), and the connection of circles marked by numbers and letters in alternating sequence (part B).
Single-task stride time | 24 weeks
  Gait will be assessed using a sensored gait mat that has embedded pressure sensors distributed throughout the mat. The mat measures location and timing of individual steps, which then can be used to calculate stride time.
Single-task stride length | 24 weeks
  Gait will be assessed using a sensored gait mat that has embedded pressure sensors distributed throughout the mat. The mat measures location and timing of individual steps, which then can be used to calculate stride length.
Single-task swing time | 24 weeks
  Gait will be assessed using a sensored gait mat that has embedded pressure sensors distributed throughout the mat. The mat measures location and timing of individual steps, which then can be used to calculate swing time.
Dual-task stride time | 24 weeks
  Gait will be assessed using a sensored gait mat that has embedded pressure sensors distributed throughout the mat. During the dual-task walking, the participants will perform 2 sets of cognitive challenges in random order: serial subtractions 3 and 5 from 100. The mat measures location and timing of individual steps, which then can be used to calculate stride time.
Dual-task stride length | 24 weeks
  Gait will be assessed using a sensored gait mat that has embedded pressure sensors distributed throughout the mat. During the dual-task walking, the participants will perform 2 sets of cognitive challenges in random order: serial subtractions 3 and 5 from 100. The mat measures location and timing of individual steps, which then can be used to calculate stride length.
Dual-task swing time | 24 weeks
  Gait will be assessed using a sensored gait mat that has embedded pressure sensors distributed throughout the mat. During the dual-task walking, the participants will perform 2 sets of cognitive challenges in random order: serial subtractions 3 and 5 from 100. The mat measures location and timing of individual steps, which then can be used to calculate swing time.
Free-living physical activity | 24 weeks
  Participants will be instructed to wear an accelerometer (GT3X+, ActiGraph, LLC) on their non-dominant wrist for 7 days. The manufacturer's software, ActiLife, will be used to process data. Physical activity counts (per minute per day over the 7 days) will be used as a measure of total physical activity.
Sleep time | 24 weeks
  Participants will be instructed to wear an accelerometer (GT3X+, ActiGraph, LLC) on their non-dominant wrist for 7 days. The manufacturer's software, ActiLife, will be used to process data to calculate total daily sleep time.
Sleep efficiency | 24 weeks
  Participants will be instructed to wear an accelerometer (GT3X+, ActiGraph, LLC) on their non-dominant wrist for 7 days. The manufacturer's software, ActiLife, will be used to process data to calculate percent sleep during in-bed intervals (sleep efficiency).

IPD SHARING:
Plan to Share IPD: No